CLINICAL TRIAL: NCT00330824
Title: Efficacy of Antibiotic Steroid Combination Compared With Individual Administration in Prevention of Post Operative Inflammation in Patients Having LASIK Surgery
Brief Title: Efficacy/Safety of Antibiotic Steroid Combination in Prevention of Post Operative Inflammation in LASIK Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Rubens Belfort Jr, Head Professor of Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BRA-05-02
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Post Lasik Surgery Inflammation
Keywords: prevention of post inflammation in LASIK surgery
MeSH Terms: interventions — Anti-Bacterial Agents; Moxifloxacin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antibiotic steroid (single vial) (Experimental): efficacy of antibiotic steroid combination compared with individual administration in prevention of postoperative inflammation in patients having LASIK surgery
  Interventions: Drug: antibiotic/steroid combination
- antibiotic / steroid (2 vials) (Active Comparator): efficacy of antibiotic steroid combination compared with individual administration in prevention of postoperative inflammation in patients having LASIK surgery
  Interventions: Drug: moxifloxacin/dexamethasone

INTERVENTIONS:
Drug: antibiotic/steroid combination — 1gtt, 4x/d, 15 days
  Other Names: moxifloxacin/dexamethasone
  Arms: antibiotic steroid (single vial)
Drug: moxifloxacin/dexamethasone — 1gtt, 4x/days, 15 days
  Other Names: moxifloxacin / dexamethasone
  Arms: antibiotic / steroid (2 vials)

SUMMARY:
Efficacy/Safety of antibiotic steroid combination compared with individual administration in inflammation Post-LASIK

DETAILED DESCRIPTION:
antibiotic/steroid combination compared to individuals components 15 days of treatment

ELIGIBILITY:
Inclusion Criteria:

* patients having LASIK surgery;
* men or women of any race, between 18 and 50 years old, presenting up to 8 degrees of myopia or up to 4 degrees of hypermetropia, or up to 3 degrees of astigmatism, without any other associated ocular problems

Exclusion Criteria:

* Uncontrolled glaucoma or intraocular hypertension;
* Use of any ocular anti-infectious drugs or any topical or systemic ocular NSAIDs during the study but study drugs;
* A history of chronic or recurrent ocular inflammatory disease;
* Uncontrolled diabetes mellitus and diabetic retinopathy ;
* Patients with sight in a single eye;
* Iris atrophy in the eye to be operated;
* Pregnant or lactating women, or women of childbearing potential who are not using proper birth-control methods;
* Known or suspected allergy or hypersensitivity to any component of study medication;
* A history or any other evidence of severe systemic disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2006-04; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
day 15 evaluation of anterior chamber | 15 days pos-op

SECONDARY OUTCOMES:
day 15 evaluation of ocular pain, physician´s follow-up impression of inflammatory reaction score | 15 days pos-op

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort Jr, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Dept. of Ophthalmology - Rua Botucatu 824, São Paulo, São Paulo, Brazil